CLINICAL TRIAL: NCT05223660
Title: A Phase 1 Single-Center Study to Assess Pharmacokinetics, Safety and Tolerability of KT07 in Healthy Adult Subjects
Brief Title: A Phase I Pharmacokinetics Study for KT07 Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yiling Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KT07-US-03
Record Dates: First submitted 2021-12-10; First posted 2022-02-04 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Healthy Adult Subjects; Pharmacokinetics; Safety and Tolerability
Keywords: Phase I; Pharmacokinetics (PK); KT07

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1 of the study is open-label. Part 2 of the study is double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose KT07 (Experimental): KT07 single dose (4 capsules) followed by multiple doses for 5 days (tid)
  Interventions: Drug: Low dose KT07
- High dose KT07 (Experimental): KT07 single dose (6 capsules) followed by multiple doses for 5 days (tid)
  Interventions: Drug: High dose KT07
- Low dose placebo (Placebo Comparator): Placebo single dose (4 capsules) followed by multiple doses for 5 days (tid)
  Interventions: Drug: Low dose Placebo
- High dose placebo (Placebo Comparator): Placebo single dose (6 capsules) followed by multiple doses for 5 days (tid)
  Interventions: Drug: High dose Placebo

INTERVENTIONS:
Drug: Low dose KT07 — A single dose of 4 capsules, followed by multiple doses on Days 8-12
  Other Names: Lianhua Qinwen
  Arms: Low dose KT07
Drug: High dose KT07 — A single dose of 6 capsules, followed by multiple doses on Days 8-12
  Other Names: Lianhua Qingwen
  Arms: High dose KT07
Drug: Low dose Placebo — A single dose of 4 capsules, followed by multiple doses on Days 8-12
  Other Names: placebo
  Arms: Low dose placebo
Drug: High dose Placebo — A single dose of 6 capsules, followed by multiple doses on Days 8-12
  Other Names: placebo
  Arms: High dose placebo

SUMMARY:
This is a phase 1 single-center study to assess the pharmacokinetics (PK), safety and tolerability of KT07 capsules in healthy adult subjects. This study consists of 2 parts: Part 1 and Part 2.

The primary objectives of Part 1 include selection of suitable PK markers for bioanalysis, development and validation of GLP bioanalytical methods for follow-up PK studies, assessment of PK of potential markers following an oral administration of KT07, and provision of PK sampling strategy for Part 2.

The primary objective of Part 2 is to evaluate the PK profile following a single dose and multiple doses in healthy adult subjects.

DETAILED DESCRIPTION:
This is a 2-part PK study. Each Part consists of 3 phases: a 2-week screening phase, drug administration and PK sampling phase, then a safety follow-up visit at Day 7 after the last dose. Subjects enter screening at Visit 1.

Part 1: Pilot single-dose PK Study Part 1 is an open-label study. Six (6) eligible male adult healthy volunteers aged between 18 to 65 years will receive a single oral dose of KT07 capsules on Day 1.

Part 2: Single and multiple-dose PK Study A total of 20 healthy subjects will participate in this part of the study, which consists of 2 cohorts with 10 subjects each. Subjects will receive either active treatment or placebo treatment in each cohort in a double-blind manner to evaluate PK and safety of KT07.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily has agreed to participate in this study and signed an Institutional Review Board (IRB)-approved informed consent before any of the screening procedures will be performed.
2. 18 to 65 years of age, inclusive, at screening, male or female.
3. Body mass index (BMI) between 17.5 and 32.0 kg/m2 at screening.
4. Healthy, determined by pre-study medical evaluation and Investigator/designee discretion (medical history, physical examination, vital signs, ECG, and clinical laboratory evaluations).
5. All female subjects of child-bearing potential must have a negative serum pregnancy test result. All female subjects of child-bearing potential and male subjects and their spouse/partner must agree to use a medically acceptable method of contraception (e.g, abstinence, an intrauterine device, a double barrier method such as condom + spermicide or condom + diaphragm with spermicide, a contraceptive implant, an oral contraceptive or have a vasectomized partner with confirmed azoospermia) throughout the entire study period, and for 90 days after study drug discontinuation.
6. Agrees to the collection of nasopharyngeal (NP) swabs for SARS-CoV-2 testing.

Exclusion Criteria:

1. Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the Investigator/designee.
2. Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
3. Any concurrent disease or condition that, in the opinion of the Investigator/designee, would make the subject unsuitable for participation in the clinical study.
4. Subject has history of alcohol and/or illicit drug abuse within one year of the Screening visit.
5. Positive SARS-CoV-2 testing by standard RT-PCR assay.
6. Positive Screening test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody.
7. Positive urine test for ethanol/drug/cotinine at Screening or Day -1.
8. History of alcohol abuse as judged by the Investigator within approximately 1 year. Average weekly alcohol intake > 21 units/week or are unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to Day -1 until completion of the study. Positive alcohol test at Screening. (One unit of alcohol equals about 250 mL of beer or lager, 100 mL of wine, or 35 mL of spirits).
9. History of illicit drug abuse, within approximately 1 year or evidence of current use as judged by the Investigator or are unwilling to abstain from illicit drug use consumption during the entire study. Positive drug test, including marijuana.
10. Excessive consumption of coffee, tea, cola, or other caffeinated beverages; excessive consumption is defined as >6 servings per day (1 serving contains approximately 120 mg caffeine).
11. Donation of blood (> 500 mL) or blood products within 2 months prior to Day -1.
12. Use of over-the-counter (OTC) vitamins and medications, prescription medications, an investigational drug or herbal remedies from 14 days prior to the first dose.
13. Subject has a history of hypersensitivity to the investigational product (IP) or any of the ingredient or excipient of IP.
14. Subjects who took a monoamine oxidase inhibitor (MAOI) within 2 weeks prior to admission.
15. Subject has consumed grapefruit or grapefruit juice within the 14 days prior to admission.
16. Pregnant or breast-feeding female subjects
17. Previous history of difficulty swallowing capsules.
18. History and/or family history of congenital long QT syndrome, unexplained syncope, or other additional risks of Torsade de Pointes or sudden premature death.
19. Subject with any of the following ECG results at Screening or Admission will be excluded:

    1. PR interval >220 msec or <110 msec
    2. RR interval > 1333 msec
    3. QRS interval >120 msec
    4. QTcF >470 msec
    5. ST segment elevation or depression considered clinically significant by the PI or designee
    6. T-wave abnormalities considered to be clinically significant by the PI or designee
20. An average systolic blood pressure ≥140 mmHg or ≤ 90 mmHg; an average diastolic blood pressure ≥ 90 mmHg or ≤ 50 mmHg.
21. Participants with history of hyperthyroidism and increased intraocular pressure.
22. Glomerular filtration rate (GFR) ≤70 mL/min/1.73 m2, as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.at Screening
23. Ongoing liver disease or unexplained liver function test (LFT) elevations, defined as alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyltransferase (GGT), or alkaline phosphatase (ALP) >1.2 × upper limit of the reference range (ULRR) at Screening or Admission
24. History of significant multiple and/or severe allergies (including latex allergy); anaphylactic reaction; or significant prescription drug, non-prescription drug, or food intolerance.
25. Any vaccination within 7 days of Screening or any vaccination with an mRNA or adenovirus platform vaccine within 30 days of Screening
26. Hemoglobin (HbA1C) > 6.5
27. Any other factors that the Investigator considers not suitable for participating in this trial.
28. Subject is unable to understand the protocol requirements, instructions and study related restrictions, as well as the nature, scope, and possible consequences of the clinical study.
29. Subject is unlikely to comply with the protocol requirements, instructions and study related restrictions, such as uncooperative attitude, inability to return for follow-up visits, and improbability of completing the clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Part 1 of the study is for male only. Part 2 of the study is for both genders.
Enrollment: 26 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) 0-t | 13 days
  AUC calculation up to the last measurable concentration
AUC0-∞ | 13 days
  AUC calculation from time 0 to infinity
Maximum (or peak) serum concentration (Cmax) | 13 days
  Assess the peak concentration of KT07
Time to achieve maximum drug concentration (Tmax) | 13 days
  Assess when KT07 reach its peak concentration
Trough concentration (Ctrough) | 13 days
  Assess the lowest concentration of KT07
Time required to reduce the drug concentration to ½ of its initial value (t1/2) | 13 days
  Assess the half-life of KT07
Volume of plasma cleared of drug per unit time (CL/F) | 13 days
  Assess the plasma clearance of KT07
Volume of distribution at terminal phase (Vz/F) | 13 days
  Assess the Volume of distribution of KT07
AUCextrap | 13 days
  Percentage of AUCinf-pred due to extrapolation from Tlast to infinity
Cmax (Racc_Cmax) | 13 days
  Maximum concentrations anticipated at plateau
AUC (Racc_AUCss) | 13 days
  Area under the curve anticipated at plateau
Accumulation factor | 13 days
  Accumulation factor (R) reflects how much drug is accumulated in the body at steady state after multiple dosing as compared to that after single dosing

SECONDARY OUTCOMES:
Severity of adverse events | 19 days
  Severity assessment of adverse events using protocol-defined criteria after first dose in adult healthy subjects
Causality of adverse events | 19 days
  Causality assessment of adverse events using protocol-defined criteria after first dose in adult healthy subjects
Incidence of adverse events | 19 days
  Incidence of adverse events up to 19 days after first dose in adult healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Nan Zhang, PhD, Study Director — Yiling Pharmaceutical
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No